CLINICAL TRIAL: NCT05871450
Title: Legacy of the Special Olympics World Games Berlin 2023
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German University of Health and Sports (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SOWG Studie
Record Dates: First submitted 2023-05-04; First posted 2023-05-23 (Actual); Results first posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Inclusion, Social
MeSH Terms: conditions — Social Inclusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants living in Host Towns (Experimental): Participants live in Host Towns, where a delegation of athletes are hosted for one week. Furthermore, Host Town coordinator organize several inclusive events.
  Interventions: Behavioral: Inclusive events
- Participants not living in Host Towns (No Intervention): Participants where no delegeation of athletes are hosted and no inclusive events are organized by Host Town coordinator.

INTERVENTIONS:
Behavioral: Inclusive events — Inclusive events such as inclusive sport festivals, citizen festivals or working groups at school are organized
  Arms: Participants living in Host Towns

SUMMARY:
This research aims to evaluate the impact of the project "170 Nations - 170 Inclusive Communities" of the Special Olympics World Games 2023 (SOWG 23) on sustain inclusive structures for people with intellectual disabilities (ID). The research utilizes a quasi-experimental research design and a qualitative research design and will synthesize qualitative and quantitative data to display successful and non-successful interventions for more inclusive communities. The research will target 56 host communities of SOWG 23 and 56 non-host communities, interviewing 200 people with ID and a minimum of 400 key stakeholders, as well as conducting qualitative interviews and focus groups.

ELIGIBILITY:
Inclusion Criteria:

* legal age

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Ruf, PhD, Study Chair — German University of Health and Sports
Locations (1):
- German University of Health and Sport, Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants Living in Host Towns | Participants Not Living in Host Towns
Started | 342 | 146
Completed | 183 | 70
Not Completed | 159 | 76

BASELINE CHARACTERISTICS:
Population: this is the toal number of participants. The difference is because some participants did not provide any information at baseline measurement.
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants Living in Host Towns | Participants Not Living in Host Towns | Total
Number analyzed (Participants) | 342 | 146 | 488
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: because participants did not provide any information
  years
    number analyzed (Participants) | 341 | 146 | 487
    (all) | 49.9 (13.1) | 52.0 (15.4) | 50.5 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants] — beca Population: because participants did not provide any information
  Participants
    Female | 159 | 69 | 228
    Male | 183 | 77 | 260
physical activity with people with intellectual disabilities [Count of Participants; unit: Participants] — Percentage of people who reported beeing physically active together with people with intellectual disabilities.
  Participants | 36 | 14 | 50
work with people with intellectual disabilities [Count of Participants; unit: Participants] — Percentage of people who stated that they work with people with intellectual disabilities.
  Participants | 111 | 51 | 162
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Attitudes Measured With the ATTID-Questionnaire
Description: The ATTID-SF Questionnaire encompassing three core components. The affective component refers to emotional responses toward individuals with intellectual disabilities. The cognitive component encompasses beliefs, knowledge, and perceptions about this population. The behavioral component reflects self-reported actions. The short form comprises 35 items rated on a 5-point Likert scale (1 = strongly agree to 5 = strongly disagree), with higher scores indicating more negative attitudes. Items are grouped into five factors: (1) interaction, (2) sensitivity/tenderness, (3) discomfort, (4) knowledge about abilities, and (5) knowledge about causes of intellectual disabilities. Mean scores are calculated for each factor; however, due to the scale's factor structure, an overall score is not recommended. So the minimum mean score for each factor is 1, the maximum means score is 5.
Time Frame: Change from baseline (T1) attitudes toward people with intellectual disability (ATTID-Questionnaire) at 3-4 month (T2) and 8-9 month (T3)
Population: The difference is due to dropouts during the follow-up assessment
Measure: Mean (Standard Deviation); unit: mean change score
Arm/Group | Participants Living in Host Towns | Participants Not Living in Host Towns
Number analyzed (Participants) | 342 | 146
mean change score
  T1 Discomfort: number analyzed (Participants) | 156 | 52
  T1 Discomfort | 1.95 (0.77) | 2.20 (0.76)
  T1 Knowledge of capacity and rights: number analyzed (Participants) | 147 | 51
  T1 Knowledge of capacity and rights | 1.78 (0.55) | 2.04 (0.55)
  T1 Interaction: number analyzed (Participants) | 142 | 48
  T1 Interaction | 2.22 (0.65) | 2.41 (0.71)
  T1 Sensitivity or tenderness: number analyzed (Participants) | 150 | 52
  T1 Sensitivity or tenderness | 2.57 (0.95) | 2.71 (0.94)
  T1 Knowledge of causes: number analyzed (Participants) | 124 | 46
  T1 Knowledge of causes | 1.89 (0.55) | 2.07 (0.42)
  T2 Discomfort: number analyzed (Participants) | 156 | 52
  T2 Discomfort | 1.92 (0.81) | 2.19 (0.76)
  T2 Knowledge of capacity and rights: number analyzed (Participants) | 147 | 51
  T2 Knowledge of capacity and rights | 1.82 (0.51) | 1.99 (0.50)
  T2 Interaction: number analyzed (Participants) | 142 | 52
  T2 Interaction | 2.21 (0.63) | 2.45 (0.64)
  T2 Sensitivity or tenderness: number analyzed (Participants) | 150 | 52
  T2 Sensitivity or tenderness | 2.57 (0.95) | 2.90 (0.91)
  T2 Knowledge of causes: number analyzed (Participants) | 124 | 46
  T2 Knowledge of causes | 1.89 (0.51) | 1.89 (0.58)
  T3 Discomfort: number analyzed (Participants) | 125 | 52
  T3 Discomfort | 1.86 (0.77) | 2.10 (0.78)
  T3 knowledge of capacity and rights: number analyzed (Participants) | 121 | 51
  T3 knowledge of capacity and rights | 1.84 (0.51) | 2.02 (0.57)
  T3 Interaction: number analyzed (Participants) | 115 | 47
  T3 Interaction | 2.22 (0.61) | 2.36 (0.72)
  T3 Sensitivity and tenderness: number analyzed (Participants) | 120 | 52
  T3 Sensitivity and tenderness | 2.65 (0.95) | 2.75 (0.89)
  T3 knowledge of causes: number analyzed (Participants) | 97 | 45
  T3 knowledge of causes | 1.81 (0.01) | 1.89 (0.63)
Statistical Analysis 1: Comparison: Participants Living in Host Towns vs Participants Not Living in Host Towns; Test type: Superiority; p = 0.05, Regression, Linear

ADVERSE EVENTS:
Time Frame: Adverse events were not monitored
Description: Adverse events were not monitored in this study because the intervention was non-invasive, low-risk, and behavioral in nature, involving only questionnaire-based assessments and/or educational or social interaction components. Based on prior literature and ethical review, the likelihood of physical or psychological harm was deemed minimal. Therefore, systematic tracking of adverse events was not considered necessary for this study design.
Arm/Group | Participants Living in Host Towns | Participants Not Living in Host Towns
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-03): https://cdn.clinicaltrials.gov/large-docs/50/NCT05871450/Prot_SAP_000.pdf